CLINICAL TRIAL: NCT03544489
Title: Clinical Effectiveness of Exercise After an ICD (E-ICD)
Brief Title: Effectiveness of Exercise After an ICD
Acronym: E-ICD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cynthia M. Dougherty, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00020647
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Heart Arrest; Implantable Defibrillator User; Physical Activity
MeSH Terms: conditions — Heart Arrest; Motor Activity

STUDY DESIGN:
Intervention Model Description: home walking exercise
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-ICD Intervention (Experimental): E-ICD Intervention over 3 months, consists of home walking to achieve the goal of 30 minutes on all or most of the days at moderate level intensity. E-ICD elements are: 1) exercise instructional DVD and manual, 2) exercise monitoring tools (Polar HR monitor, Borg scale, and exercise logs), and 3) telephone coaching by cardiac rehabilitation (CR) staff. Each participant receives an exercise prescription based on the ICD information using HR cut-offs, a minimum of 4 walking sessions/week will be prescribed. Exercise maintenance: At the 3 month conclusion of the E-ICD intervention, each patient will receive an exercise prescription based on the level they were able to achieve, with guidelines about increasing exercise to reach the target of 30 minutes/walking on all or most days over the ensuing 3 months.
  Interventions: Behavioral: E-ICD Intervention
- Usual Care (No Intervention): Usual Care will receive treatment "as usual" from their health care clinicians with outcomes measured at baseline, 3, 6, and 12 months. Participants will not be discouraged from physical activity, but will be asked not to change their current level of activity for 6 months while in the study. Usual care involves ICD interrogation and follow-up every 3 months, measured either in-person or with home telephonic transmissions. Because participants in usual care may choose to participate in another exercise program, we will monitor those who participate in exercise programs and use the StepWatch monitor to quantify the amount and timing of physical activity. To control for group differences in attention, investigators will telephone usual care participants requesting information about health care utilization twice during the study at 3, 6, and 12 months.

INTERVENTIONS:
Behavioral: E-ICD Intervention — Home walking 3 days/week x 12 weeks
  Arms: E-ICD Intervention

SUMMARY:
This study will test an exercise intervention (E-ICD) following an implantable cardioverter defibrillator.

DETAILED DESCRIPTION:
The goal of this study is to test the effectiveness and describe implementation of a home based exercise intervention for persons with an implantable cardioverter defibrillator (ICD). This study is based on the NIH stage model of behavioral interventions (stage III effectiveness) that aligns with the strategic mission of the NHLBI, to optimize clinical and implementation research to improve health and reduce disease (Obj #6). The study intervention is based on the protocol and monitoring components that were developed in prior RCTs and a pilot study conducted by our team. From these studies, we created a home based exercise program called Exercise-ICD (E-ICD) for testing in a broader range of ICD patients, that assists individuals to start and monitor exercise safely after an ICD. An randomized two group (E-ICD vs. usual care) pragmatic effectiveness mixed-methods study is proposed, to determine the effectiveness of the E-ICD intervention and describe implementation by cardiac rehabilitation (CR) clinical staff. Two hundred ten (N=210) patients in 3 local study sites (70/site) in the greater Seattle, WA area will participate. E-ICD is guided by the Reach-Effectiveness-Adoption-Implementation-Maintenance (RE-AIM) model. The E-ICD intervention consists of 12 weeks of home walking exercise using exercise prescriptions and protocols validated in our previous work. The primary effectiveness outcome is patient physical activity (steps/day) after the E-ICD intervention at 3 months. We will determine the number of patients who reach the public health walking goal of moderate level exercise of 150 minutes/week at the end of the study. Measures will be taken at baseline, after the intervention at 3 months, and at 6 and 12 months to determine maintenance. The specific aims are to: 1) Test the hypothesis that participants randomized to E-ICD vs. usual care (UC) will demonstrate increased physical activity (minutes walked/week) [primary outcome], health related quality of life, gait speed, mobility, exercise self-efficacy; and reduced ICD shock anxiety and depression at 3 months (E-ICD Effectiveness), 2) Assess longer term effects of E-ICD on participant and health care system Maintenance, captured by 1) participant retention, satisfaction, and adherence at 12 months (total minutes/week), and 2) clinician and institutional intent to sustain use of the E-ICD intervention after the study, and 3) Evaluate the reach, adoption, and implementation of E-ICD by CR clinical staff. Reach will be assessed by the diverse patient participation rate, representativeness, and reasons for non-interest. Adoption is the participation rate and representativeness of the settings and staff who participate, and factors related to adoption. Implementation will be assessed by delivery fidelity of E-ICD and workflow adaptations, implementation costs, and consistency of delivery across settings.

ELIGIBILITY:
Inclusion Criteria:

* ICD implantation for primary or secondary prevention of sudden cardiac arrest, -ability to read, speak and write English,-
* access to a reliable phone for 6 months after study entry,
* able to ambulate without assist devices for at least 5-10 minutes/day
* greater than 18 years of age.

Exclusion Criteria:

* current diagnosis of serious mental disorder,
* regular non-medical use of illicit drugs (opiates, cocaine, amphetamines, etc.), -unstable angina, myocardial infarction, ICD shock or heart surgery within previous 3 months
* pregnancy
* concurrent participation in an exercise program > 5 days/week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-09-14 (Estimated); Study Completion 2029-09-14 (Estimated)

PRIMARY OUTCOMES:
Daily activity | Baseline, 3, 6, and 12 months
  average steps/day measured on Step Watch activity monitor

SECONDARY OUTCOMES:
General Health | Baseline, 3, 6, and 12 months
  PROMIS Global v1.2 measures 5 domains of global health and quality of life, including physical, mental, and social health. Two factors physical health (GPH) and mental health (GMH) are derived.
Mobility | Baseline, 3, 6, and 12 months
  PROMIS Mobility V2.1 measures general mobility of lower extremities in adults, relating to overall physical functioning
Self-Efficacy for Walking | Baseline, 3, 6, and 12 months
  Self-Efficacy for Exercise Scale (9-items, α=0.92) assesses self-efficacy expectations related to one's ability to walk in the face of barriers to exercise [22], was used in the pilot and found to be sensitive to change with the intervention.
ICD shock anxiety | Baseline, 3, 6, and 12 months
  Florida Shock Anxiety Scale (FSAS), assesses anxiety about receiving an ICD shock [23], is sensitive to change across time.
Depression | Baseline, 3, 6, and 12 months
  Patient Health Questionnaire-9 (PHQ-9) (9 items, α=0.83), measures depressive symptoms, as well as suicidality.

OTHER OUTCOMES:
Long Term Maintenance | 12 months
  Measure of innovation-specific implementation intentions (MISII) scale (3 items) completed by CR staffs and site staff, measures the providers' intentions to use the E-ICD program in routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Dougherty, ARNP, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No